CLINICAL TRIAL: NCT03033056
Title: Neurobiology of Generalized Fear-Conditioning & Avoidance in Anxiety Disorders (Community Anxiety Response Study)
Brief Title: Neurobiology of Generalized Fear-Conditioning & Avoidance in Anxiety Disorders
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1610M96641
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anxiety Disorders
Keywords: fear-conditioning; behavioral avoidance; anxiety disorders; fMRI
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anxiety Clinic Patients: Adult males and females being treated at the anxiety disorders clinic at the University of Minnesota predominantly for clinical anxiety.
  Interventions: Behavioral: Test of fear conditioning
- Healthy Comparisons: Sex, age, and socioeconomically matched healthy controls
  Interventions: Behavioral: Test of fear conditioning

INTERVENTIONS:
Behavioral: Test of fear conditioning — Behavioral and brain correlates of conditioned fear generalization and avoidance will be assessed using fMRI and related to levels of anxiety related psychopathology.

SUMMARY:
Anxiety disorders are among the most prevalent, costly, and disabling mental illnesses. One central, yet largely understudied, abnormality in anxiety disorders is the heightened tendency to display fear and avoidance in reaction to benign or safe events that resemble feared situations. The current project maps brain circuits associated with this abnormality in order to contribute to future brain-based diagnosis and treatments for clinical anxiety.

DETAILED DESCRIPTION:
The objective of this project is to neurally, behaviorally, psychologically, and clinically characterize fundamental Pavlovian and instrumental dimensions of potential threat through which emotional and behavioral responses to threat cues generalize to resembling, safe stimuli. Such generalization is aligned with the potential threat construct due to the threat ambiguity, or uncertain threat value, inherent in these safe 'generalization' stimuli. The Pavlovian dimension of interest is generalization of conditioned fear: a fundamental Pavlovian process through which fear transfers, or generalizes, to safe stimuli resembling a conditioned threat-cue (CS+). The targeted instrumental dimension is generalized avoidance: active decisions to withdraw from safe stimuli resembling the CS+ that are motivationally prompted by Pavlovian generalization. Given lab-based findings have linked heightened Pavlovian generalization to a variety of traditional anxiety disorders, overgeneralization represents a promising dimension of potential threat with relevance across traditional anxiety disorders. One central aspect of this project is testing personality and psychiatric factors (e.g., trait fear, internalizing, externalizing) that may account for the relevance of generalization and its neurobiology across traditional anxiety disorders. A second key aspect, is studying neural processes by which Pavlovian generalization evokes instrumental generalized avoidance of benign stimuli (resembling danger cues), which, when excessive, is likely to impair day-to-day functioning in anxiety patients. Unfortunately, human fear-conditioning experiments in clinical samples, have focused almost exclusively on passive-emotional, Pavlovian conditioning, to the virtual exclusion of studying active-behavioral, instrumental avoidance. The current neuroimaging project fills this gap by applying a novel Pavlovian-instrumental generalization paradigm to neurally and behaviorally elucidate Pavlovian processes leading to generalized instrumental avoidance. Personality moderators (e.g., dispositional resilience) of relations between Pavlovian and instrumental generalization will also be examined. The studied adult samples will display a wide range of symptom severity across traditional anxiety disorders and will include anxiety-clinic patients and healthy comparisons (N=159). Central goals of this proposal include: 1) elucidating the neurobiology of Pavlovian and instrumental generalization and their interaction, 2) testing relations between neural substrates of Pavlovian and instrumental generalization and broad psychiatric dysfunction (Aims2-3); and 3) assessing the degree to which relations between these dimensions of generalization and broad dysfunction are driven by psychometrically validated personality traits relevant across traditional anxiety disorders. This third and final goal is critical to the project, because individual difference measures capturing empirically-validated psychological constructs will likely track relations between fundamental conditioning processes (e.g., generalization) and general dysfunction, better than traditional, polythetic, diagnostic entities, that, by and large, do not reflect any single coherent psychological process.

ELIGIBILITY:
Inclusion Criteria:

A. Diagnosis: No psychiatric diagnosis is required, but recruitment will be guided by the goal of attaining a sample with wide-ranging levels of both anxiety symptom severity and individual differences in anxiety-related states and traits.

B. Caffeine and tobacco use: Participants will abstain from caffeine and tobacco one hour preceding testing

Exclusion Criteria:

A. Psychiatric health: Current or past history of any psychotic disorder, bipolar disorder, delirium, dementia, amnestic disorder, or mental retardation; comorbid depression if accompanied by current, significant suicide risk; substance use disorder presently or for the six months preceding testing.

B. Current use of any medication that alters central nervous system function including antidepressants, benzodiazepines, anti-psychotics, mood stabilizers,anti-parkinsonian agents, anti-convulsants, sleep medications, pain medications, and anti-hypertensives.

C. Medical health: Current or past medical illnesses which in the investigator's opinion may confound study results, or place the participant at risk.

D. Pregnancy status: Females who are, or may be, pregnant. Recruitment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female adults presenting with anxiety symptoms at the Anxiety Disorders Clinic in the Department of Psychiatry at U of MN, as well as demographically matched healthy comparisons
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging | Years 1-4
  Blood oxygenation level dependent responses elicited during the fear conditioning paradigm

SECONDARY OUTCOMES:
Behavioral measures | Years 1-4
  Online behavioral responses elicited during the fear conditioning paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Lissek, PhD, Principal Investigator — U of MN
Locations (1):
- University of MInnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No